CLINICAL TRIAL: NCT02860351
Title: The Effect of Head Positioning on the Cross-sectional Area of the Subclavian Vein
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, M.D, SMG-SNU Boramae Medical Center
Other Study IDs: PRE20160711-001
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Normal Volunteers
Keywords: subclavian vein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the present study, the cross-sectional area of subclavian vein, the distances of subclavian vein ~ subclavian artery and subclavian vein ~ pleura are assessed in different head positions (neutral, rotation to ipsilateral or contralateral sides) in spontaneous breathing adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Medication affecting vascular elasticity
* History of central venous catheterization or clavicle fracture
* History of lung surgery, operation of chest cage

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults ≥ 20 yr
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-08-10; Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of subclavian vein | through study completion, an average of 1 year

SECONDARY OUTCOMES:
depth of subclavian vein from skin | through study completion, an average of 1 year
Distance of subclavian vein ~ subclavian artery | through study completion, an average of 1 year
Distance of subclavian vein ~ pleura | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Chang JE, Lee JM, Han SH, Ryu JH, Hwang JY. The Effect of Head Position on the Cross-Sectional Area of the Subclavian Vein. Anesth Analg. 2018 Jun;126(6):1946-1948. doi: 10.1213/ANE.0000000000002446. PMID 28863021